CLINICAL TRIAL: NCT00460512
Title: An Open-label Prospective Trial to Explore the Tolerability, Safety and Efficacy of Flexibly Dosed Paliperidone ER in Subjects With Schizophrenia
Brief Title: An Efficacy, Safety And Tolerability Study of Flexibly Dosed Paliperidone Extended Release (ER) in Participants With Schizophrenia
Acronym: PERFlexS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR012949; R076477SCH3017 (Other: Janssen-Cilag International NV); 2006-004265-34 (EudraCT Number)
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Flexible dosing; Non-acute patients; Antipsychotic; Atypical; INVEGA
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Paliperidone Extended Release (ER) (Experimental)
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — Paliperidone ER tablet in dose range of 3 to12 milligram (mg) per day was given orally for 6 months as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics due to lack of efficacy, lack of tolerability, lack of compliance or other reasons.

SUMMARY:
The purpose of this study is to explore tolerability, safety and effectiveness of flexibly dosed paliperidone extended release (ER) in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) previously unsuccessfully treated with an oral antipsychotic medication.

DETAILED DESCRIPTION:
This is a non-randomized (the study drug is not assigned by chance), single arm, multicenter (when more than one hospital or medical school team work on a medical research study) 6-month study. Participants can be transitioned to an effective dose of paliperidone ER from any oral antipsychotic medication due to lack of efficacy, lack of tolerability or safety, lack of compliance or other reason. A transition period of maximum 4 weeks will be allowed. Throughout the study, participants will receive flexible dose of 3 to 12 milligram (mg) of paliperidone once daily orally for 6 months. Adjustment of the dosage will be done at Investigator's discretion, based on the individual participant's clinical response and tolerability of the study drug dosages. Participants who complete this 6-month study and would like to continue will be eligible to be enrolled in an extension phase until paliperidone ER is available. The starting dose of the extension phase will be the same as at the end of the 6-month study and may be changed throughout the extension period. The extension phase will consist of a main extension phase (ending with an End of Main Extension Phase Visit) and a modified extension phase (ending with an End of Study Visit). Efficacy will primarily be evaluated by positive and negative syndrome scale (PANSS). Safety will primarily be evaluated by Extrapyramidal Symptom Rating Scale (ESRS).

ELIGIBILITY:
Inclusion Criteria:

* Participant meets the Diagnostic and Statistical Manual of Mental Disorders (Edition 4) criteria for schizophrenia
* Participant is previously non-acute (on the same antipsychotic medication used for the treatment of schizophrenia and Clinical Global Impression-Severity [CGI-S] change less than or equal to 1 in the past 4 weeks before enrollment) and has been given an adequate dose of an appropriate oral antipsychotic for an adequate period of time prior to enrollment, but previous treatment is considered unsuccessful due to one or more of the following reasons: lack of effectiveness, lack of tolerability or safety, lack of compliance and/or other reasons to switch to another antipsychotic medication
* Participant is healthy on the basis of a physical examination and vital signs at screening
* Female participants must be postmenopausal for at least 1 year, surgically sterile, abstinent, or, if sexually active, agree to practice an effective method of birth control before entry and throughout the study
* Participants must be willing and able to fill out self-administered questionnaires

Exclusion Criteria:

* Participants on clozapine, any conventional depot neuroleptic or risperidone long-acting injection during the last 3 months
* Participants with serious unstable medical condition, including known clinically relevant laboratory abnormalities
* Participants with history or current symptoms of tardive dyskinesia (twitching or jerking movements that you cannot control in your face, tongue, or other parts of your body) and neuroleptic malignant syndrome (high fever, rigid muscles, shaking, confusion, sweating more than usual, increased heart rate or blood pressure, or muscle pain or weakness)
* Participants judged to be at high risk for adverse events, violence or self-harm
* Participants with a current use or known history (over the past 6 months) of substance dependence according to Diagnostic and Statistical Manual of Mental Disorders (Edition 4) Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1814 (Actual)
Dates: Start 2007-04-25 (Actual); Primary Completion 2009-01-22 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With at Least 20 Percent Improvement in Total Positive and Negative Syndrome Scale (PANSS) Score in Those Participants who Transitioned due to Lack of Efficacy | Endpoint (up to Week 26)
  The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self). The PANSS provides a total score and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each item scored on a scale of 1 (absent) to 7 (extreme). The total score ranges from 30 to 210 and higher score indicates greater severity.
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Endpoint (up to Week 26) | Baseline and endpoint (up to Week 26)
  The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia. The PANSS provides a total score and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each item scored on a scale of 1 (absent) to 7 (extreme). The total score ranges from 30 to 210 and higher score indicates greater severity.

SECONDARY OUTCOMES:
Percentage of Participants With at Least 20 Percent Improvement in Total Positive and Negative Syndrome Scale (PANSS) Score | Endpoint (up to Week 26)
  The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self). The PANSS provides a total score and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each item scored on a scale of 1 (absent) to 7 (extreme). The total score ranges from 30 to 210 and higher score indicates greater severity.
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Subscale Scores at Endpoint (up to Week 26) | Baseline and endpoint (up to Week 26)
  The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia. The PANSS provides a total score and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each item scored on a scale of 1 (absent) to 7 (extreme). Positive subscale score ranges from 7 (absent) to 49 (extreme psychopathology), negative subscale score ranges from 7 (absent) to 49 (extreme psychopathology) and general psychopathology subscale score ranges from 16 (absent) to 112 (extreme psychopathology).
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Marder Subscale Scores at Endpoint (up to Week 26) | Baseline and endpoint (up to Week 26)
  The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). Marder PANSS subscales include positive symptoms subscale consisting of 8 items with total score range of 8-56; negative symptoms subscale and disorganized thoughts subscale, each consisting of 7 items with total score range of 7-49; and uncontrolled hostility/excitement subscale and anxiety/depression subscale, each consisting of 4 items with total score range of 4-28. Higher score indicates greater severity.
Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score at Endpoint (up to Week 26) | Baseline and endpoint (up to Week 26)
  The CGI-S rating scale assesses the severity of a participant's psychotic condition on a 7-point scale ranging from 1 (not ill) to 7 (extremely severe).
Change From Baseline in Total Personal and Social Performance (PSP) Score at Endpoint (up to Week 26) | Baseline and endpoint (up to Week 26)
  The PSP scale assesses the degree of dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care and disturbing and aggressive behavior. The score ranges from 1 to 100, divided into 10 equal intervals to rate the degree of difficulty (1, absent to 6, very severe) in each of the 4 domains. Participants with a score of 71 to 100 have a mild degree of difficulty; from 31 to 70, varying degrees of disability; less or equal to 30, functioning so poorly as to require intensive supervision.
Change From Baseline in Short-Form 36 Health Survey (SF-36) Score at Endpoint (up to Week 26) | Baseline and endpoint (up to Week 26)
  The SF-36 is a health status survey with 36 questions measuring 8 dimensions (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health) that are subsequently aggregated into 2 summary scales, Physical Component Summary (PCS) and Mental Component Summary (MCS). Each item is scored into on a 0-100 range so that the lowest and highest possible scores are set at 0 and 100, respectively. All items are scored so that a high score defines a more favorable health state.
Number of Participants With Satisfaction With the Study Treatment | Endpoint (up to Week 26)
  Participants will assess their satisfaction with paliperidone ER on a 5-point scale: 1 (very good), 2 (good), 3 (moderate), 4 (poor) and 5 (very poor).
Change From Baseline in Sleep and Daytime Drowsiness Evaluation Score at Endpoint (up to Week 26) | Baseline and endpoint (up to Week 26)
  The Sleep and Daytime Drowsiness Evaluation Scale is a self-administered scale that rates quality of sleep and daytime drowsiness. Participants indicate on an 11 point scale how well they have slept in the previous 7 days, score ranging from 0 (very badly) to 10 (very well) and how often they have felt drowsy within the previous 7 days, score ranging from 0 (not at all) to 10 (all the time).
Change From Baseline in Extrapyramidal Symptoms Rating Scale (ESRS) Total Score at Endpoint (up to Week 26) | Baseline and endpoint (up to Week 26)
  The ESRS scale assesses parkinsonism (slow movements), dystonia (abnormal muscle movement causing focal/generalized, sustained muscle contractions, postures, and involuntary movements) and dyskinetic (involuntary muscle contractions) movement subscale. Parkinsonism consists of 8 items rated on a 7-point scale (0=absent/normal and 6=worst score), Dystonia consists of 2 items rated on a 7-point scale (0=absent and 6=extremely severe) and Dyskinetic movements consists of 7 items rated on a 7-point scale (0=none and 6=worst score). Total score: 0-102. Lower scores indicate better condition.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (231):
- Belgium (15):
  - Antwerp
  - Bertrix
  - Dave
  - Diest
  - Duffel
  - Kortenberg
  - Liège
  - Montignies-sur-Sambre
  - Mortsel
  - Roeselare
  - Saint Denijs-Westrem
  - Saint-Servais
  - Sint-Truiden
  - Tielt
  - Waregem
- Bulgaria (3):
  - Bulgaria
  - Sofia
  - Tzerova Korya
- Croatia (4):
  - Osijek
  - Rijeka
  - Split
  - Zagreb
- Denmark (4):
  - Aalborg
  - Elsinore
  - Risskov
  - Viby J
- Finland (4):
  - Ekenäs
  - Helsinki
  - Raahe
  - Tampere
- France (25):
  - Bar-le-Duc
  - Bordeaux
  - Bourg-en-Bresse
  - Bully-les-Mines
  - Caen
  - Chambéry
  - Clermont-Ferrand
  - Créteil
  - Dijon
  - Dole
  - Henin Baumont
  - Jarnac
  - La Roche-sur-Yon
  - La Seyne-sur-Mer
  - Mont-Saint-Martin
  - Montpellier
  - Nîmes
  - Paris
  - Pau
  - Rennes
  - Roubaix
  - Saint-Avé
  - Saint-Cyr-au-Mont-d'Or
  - Saint-Germain-en-Laye
  - Villejuif
- Germany (73):
  - Aalen
  - Achim
  - Augsburg
  - Bamberg
  - Bergfelde
  - Bergheim
  - Berlin
  - Bochum
  - Butzbach
  - Chemnitz
  - Coesfeld
  - Cologne
  - Darmstadt
  - Dillingen
  - Dresden
  - Duisburg
  - Düsseldorf
  - Ebensfeld
  - Eberbach
  - Ellwangen
  - Elmshorn
  - Essen
  - Ettlingen
  - Freiburg im Breisgau
  - Gelnhausen
  - Gelsenkirchen
  - Giessen
  - Göttingen
  - Haina
  - Halle
  - Hamburg
  - Hanover
  - Hattingen
  - Hemer
  - Hemmoor
  - Heppenheim an der Bergstrasse
  - Idar-Oberstein
  - Jena
  - Kaufbeuren
  - Königsbrück
  - Krefeld
  - Leipzig
  - Liebenburg
  - Lüdenscheid
  - Mainz
  - Mannheim
  - Mittweida
  - München
  - Münster
  - Naumburg
  - Norden
  - Nuremberg
  - Ober-Ramstadt
  - Oldenburg
  - Oranienburg
  - Ostfildern
  - Potsdam
  - Rostock
  - Saalfeld
  - Salzgitter
  - Schlüchtern
  - Siegen
  - Spremberg
  - Stralsund
  - Straubing
  - Ulm
  - Viersen
  - Wasserburg
  - Wiesbaden
  - Wiesloch
  - Wilhelmshaven
  - Wismar
  - Würzburg
- Greece (5):
  - Athens
  - Chios
  - Heraklion
  - Larissa
  - Thessalonikis
- Hungary (4):
  - Balassagyarmat
  - Budapest
  - Kecskemét
  - Sopron
- Israel (4):
  - Bat Yam
  - Be'er Ya'acov
  - Jerusalem
  - Pardesiyya
- Latvia (5):
  - Daugavpils
  - Jelgava
  - Liepāja
  - Riga
  - Strenči
- Lithuania (3):
  - Kaunas
  - Panevezys
  - Vilnius
- Netherlands (10):
  - Assen
  - Beilen
  - Bennebroek
  - Enschede
  - Groningen
  - Hoofddorp
  - Leeuwarden
  - The Hague
  - Tilburg
  - Zwolle
- Poland (5):
  - Bydgoszcz
  - Gdynia Na
  - Krakow Na
  - Lubliniec
  - Skorzewo Na
- Portugal (6):
  - Angra do Heroísmo
  - Braga
  - Castelo Viegas
  - Coimbra
  - Lisbon
  - Porto
- Russia (8):
  - Kazan'
  - Krasnodar
  - Moscow
  - Moscow Russia
  - Saint Peterburg Na
  - Saint Petersburg
  - Saratov
  - Yaroslavl
- Serbia (3):
  - Belgrade
  - Kragujevac
  - Novi Sad
- Spain (10):
  - Alicante
  - Barcelona
  - Bunyola Illes Balears
  - Burgos
  - Oviedo
  - Pontevedra
  - Sama de Langreo Asturias
  - Valencia
  - Zamora
  - Zaragoza
- Sweden (13):
  - Bromma
  - Gothenburg
  - Hudiksvall
  - Karlskrona
  - Malmo
  - Mölndal
  - Norrtälje
  - Nyköping
  - Simrishamn
  - Skövde
  - Solna
  - Trollhättan
  - Västra Frölunda
- Switzerland (16):
  - Aarau
  - Basel
  - Basel Bs
  - Biel/Bienne
  - Geneva
  - Lenzburg
  - Liestal
  - Marsens
  - Montreux
  - Münsingen
  - Oetwil
  - Riehen
  - Sarnen
  - Solothurn
  - Viganello
  - Zurich
- Turkey (Türkiye) (5):
  - Ankara
  - Denizli
  - Diyarbakır
  - Gaziantep
  - Izmir
- United Kingdom (6):
  - Barnet
  - Birmingham
  - Clacton-on-Sea
  - Devon
  - Exeter
  - Glasgow

REFERENCES:
- [Result] Schreiner A, Lahaye M, Peuskens J, Naber D, Dilbaz N, Millet B, Franco MA, Rancans E, Turczynski J, Smeraldi E, Lara E, Neznanov NG. Paliperidone extended-release in patients with non-acute schizophrenia previously unsuccessfully treated with other oral antipsychotics. Expert Opin Pharmacother. 2014 Apr;15(5):593-603. doi: 10.1517/14656566.2014.884071. Epub 2014 Feb 3. PMID 24491033